CLINICAL TRIAL: NCT06410144
Title: Improving Kidney Therapy Decision-Making for Older People With Advanced Chronic Kidney Disease (CKD)
Brief Title: Chronic Kidney Disease-Education (CKD-EDU)
Acronym: CKD-EDU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Fahad Saeed, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00009330; R01AG082891 (NIH)
Record Dates: First submitted 2024-05-02; First posted 2024-05-13 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Medicare Part A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research coordinators responsible for administering assessments will remain blinded to the patient's randomization status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Program A (Active Comparator): Kidney therapy education and support with kidney therapy educator.
  Interventions: Behavioral: Program A
- Program B (Active Comparator): Behavioral: CKD-EDU Palliative care-based decision-support intervention for support with kidney therapy decision-making.
  Interventions: Behavioral: Program B

INTERVENTIONS:
Behavioral: Program A — Subjects in the Control group will receive 1) National Kidney Foundation information, and 2) support from a kidney therapy educator.
  Arms: Program A
Behavioral: Program B — Subjects in the intervention group will receive 1) a video and paper decision aid, and 2) coaching from a decision support specialist. The visits will be aimed at supporting patients with kidney therapy decision-making.
  Other Names: CKD-EDU Intervention
  Arms: Program B

SUMMARY:
The investigators are conducting a study to see which program better helps older patients with kidney disease choose their treatment. Investigators are also investigating if either program can reduce the number of hospital or emergency room visits in the first 6 months of the study, as well as potentially improve end-of-life care for older adults.

Half of the participants will receive Program A, while the other half will receive Program B. Investigators will compare the two groups to see which participants feel better prepared about their kidney therapy decisions, experience improved end-of-life care, and have fewer emergency room visits and hospital admissions.

Participants in Program A will receive information from the National Kidney Foundation and meet with a kidney therapy educator. Participants in Program B will get information about kidney disease treatment and meet with a decision-support specialist who's an expert in decision-making.

DETAILED DESCRIPTION:
Older adults ≥75 years represent the fastest-growing population to initiate dialysis in the US; despite the life-altering effects of dialysis on quality of life, dialysis is often presented as a default without considering patient preferences, prognosis, and alternative options such as conservative kidney management. This study will test the first palliative care intervention for older patients with advanced chronic kidney disease to improve the kidney therapy decision-making process. This research not only has the potential to help thousands of older patients with advanced chronic kidney disease who often have unanswered questions, unmet information needs, and restricted opportunities to share personal treatment preferences with their nephrologists but also has the possibility of creating new models of collaborative care by integrating palliative care into routine nephrology care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years old
* Has advanced kidney disease with kidney function less than 30%
* Speaks English
* Has not yet made a dialysis decision

Exclusion Criteria:

* Has already decided on dialysis or active medical care without dialysis.
* Has already been seen by a Palliative Care (PC) clinician for kidney-related issues or is enrolled in hospice
* Currently on dialysis
* Unable to provide informed consent or complete verbally administered surveys due to health, sensory, or cognitive impairment.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Changes in Kidney Therapy Decision-Making Process using the Decisional Conflict Scale at 12 weeks | Baseline, 4-6 weeks, and 12 weeks
  Determine whether the intervention improves kidney therapy decision-making at 12 weeks by using the Decisional Conflict Scale. Score ranges from 0-100. Lower scores indicate better outcomes.

SECONDARY OUTCOMES:
Changes in patients' well-being at 6 months using the Burden of Kidney Disease Subscale | Base line 6 months
  Determine whether the intervention improves patient well-being at 6 months using the Burden of Kidney Disease Subscale, a 4-question scale with response options ranging from 'definitely true (0)' to 'definitely false (3)'. Higher scores indicate better outcomes.
Changes in number of hospital admissions, intensive care admissions, and emergency room visits | Baseline, 6 months
  Review electronic health records to determine whether the intervention reduces the number of hospital admissions, intensive care admissions, and emergency room visits between study entry and 6 months.
Differences in end-of-life care between intervention and control arm | Baseline to 6 months
  Review patients' medical charts to determine whether the intervention improves end-of-life care treatment during the last 30 days of life, as measured by the rates of aggressive procedures such as cardiopulmonary resuscitation (CPR), dialysis, intubation, gastrostomy (G-tube), etc.

CONTACTS AND LOCATIONS:
Overall Officials: Fahad Saeed, MBBS, MSCI, Principal Investigator — University of Rochester
Locations (5):
- United States (5):
  - UR Medicine Nephrology - Strong West, Brockport, New York
  - Nephrology Clinic - Thompson Professional Building, Canandaigua, New York
  - Nephrology Clinic - St. James Medical Office Building, Hornell, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified qualitative data will be available to other researchers.